CLINICAL TRIAL: NCT00184093
Title: Phase I/II Study of Gemcitabine and Concurrent Radiation Followed by Adjuvant Hysterectomy in Bulky Stage Ib and IIa Cervical Carcinoma: Analysis of Prognostic Factors and Determinants of Response: A Pilot Study
Brief Title: Study of Gemcitabine and Concurrent Radiation Followed by Adjuvant Hysterectomy in Bulky Stage Ib and IIa Cervical Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5C-99-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Uterine Cervical Cancer
Keywords: Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Gemcitabine

ARMS (1):
- Gemcitabine weekly x 6 wks with concurrent external radiation (Experimental): Gemcitabine 350 mg/m2 IV weekly x 6 weeks with concurrent external radiation
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine weekly x 6 wks with concurrent external radiation

SUMMARY:
The purpose of this study is first to establish what is the ideal dose of gemcitabine, a chemotherapy agent, when given in combination with radiation. In addition, the investigators want to determine the side effects and the effectiveness of this combination. The investigators will also study several markers to try to identify markers or tests that will predict which patients will benefit more from this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed bulky stage Ib or stage IIa cervical cancer. Bulky stage Ib disease is defined as tumor mass greater than 4 cms in diameter.
* Cervical lesion which is measurable by physical examination.
* No prior therapy for invasive cervical cancer.
* GOG performance status 0-2
* Signed informed consent
* Patients must have adequate:

  * Bone marrow function: absolute granulocyte count > or = to 1500, platelet count > 100,000.
  * Renal function: creatinine < or = to 1.8 mg/dl
  * Hepatic function: bilirubin < or = to 1.5 x normal, SGOT and alkaline phosphatase < or = to 3 x normal

Exclusion Criteria:

* Patients with a history of prior malignancy, except adequately treated basal cell or squamous cell carcinoma of the skin, or other cancer for which the patient has been disease free for at least five years.
* Pregnant or lactating women. Women of reproductive age may not participate unless they have agreed to use an effective method of birth control.
* Patients with uncontrolled infection.
* Patients who are HIV positive
* Patients with psychiatric or social conditions that would interfere with consent or follow-up.
* Patients with any other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 1999-06; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Roman, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began recruiting in July 1999 and recruitment ended in May 2008. All participants were seen and treated at USC Norris Comprehensive Cancer Center and/or at LAC+USC Medical Center.
Pre-assignment Details: The study had no pre-assignment criteria. This was an open label study and all participants were given the same treatment.
Period: Overall Study
Arm/Group | Gemcitabine Weekly x 6 Wks With Concurrent External Radiation
Started | 35 (Phase 1 participants = 6 Phase 2 participants = 29)
Completed | 26
Not Completed | 9
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine Weekly x 6 Wks With Concurrent External Radiation
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 33
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Toxicity (Number of Participants With Serious Adverse Events)
Description: Summary of grade 3 or higher toxicities as per Common Toxicity Criteria version 2.0. Phase 1 and 2 Combined (N=35)
Time Frame: Every 3 weeks from start of study until 30 days after the last dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine Weekly x 6 Wks With Concurrent External Radiation
Number analyzed (Participants) | 35
Participants | 10

2. Secondary Outcome: Best Overall Response of Either a Complete Response (CR) or Partial Response (PR)
Description: Participants who complete the 6 weeks of chemotherapy and radiation or who experience dose limiting toxicity or who progress at any time prior to completion of the 6 weeks of chemotherapy and radiation will be evaluable for response.
  Complete response (CR): Complete disappearance of all measurable and evaluable disease. No new lesions. No disease related symptoms. No evidence of nonevaluable disease, including normalization of markers and other abnormal lab values. All measurable, evaluable, and nonevaluable lesions and sites must be assessed using the same technique as baseline.
  Partial response (PR): Applies only to patients with at least one measurable lesion. Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions. All measurable and evaluable lesions and sites must be assessed using the same techniques as baseline.
Time Frame: Baseline to response (up to 24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine Weekly x 6 Wks With Concurrent External Radiation
Number analyzed (Participants) | 35
Participants | 32

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning cycle 1 and continued throughout the study until 30 days after the last dose.
Arm/Group | Gemcitabine Weekly x 6 Wks With Concurrent External Radiation
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 10/35
Other Adverse Events (participants affected / at risk) | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine Weekly x 6 Wks With Concurrent External Radiation (N=35)
Alkaline phosphatase (Hepatobiliary disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 10 (14)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6 (6)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 (5)
Proctitis (Gastrointestinal disorders) | 2 (2)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 1 (1)
Rectal or perirectal pain (proctalgia) (General disorders) | 1 (1)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 2 (2)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 5 (6)
Vaginal bleeding (Reproductive system and breast disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine Weekly x 6 Wks With Concurrent External Radiation (N=35)
Abdominal pain or cramping (Gastrointestinal disorders) | 17 (25)
Alkaline phosphatase (Hepatobiliary disorders) | 12 (16)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Anorexia (Gastrointestinal disorders) | 27 (44)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 4 (5)
Auditory/Hearing-Other (not specified) (Ear and labyrinth disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 24 (35)
Constitutional Symptoms-Other (not specified) (General disorders) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Creatinine (Renal and urinary disorders) | 1 (1)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 33 (67)
Dizziness/lightheadedness (Nervous system disorders) | 15 (23)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dysuria (painful urination) (Renal and urinary disorders) | 28 (44)
Edema (General disorders) | 6 (9)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 23 (51)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 5 (6)
Headache (Nervous system disorders) | 22 (36)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 24 (50)
Hot flashes/flushes (Endocrine disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (8)
Hypoalbuminemia (Hepatobiliary disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 10 (10)
Inner ear/hearing (Ear and labyrinth disorders) | 5 (11)
Insomnia (Psychiatric disorders) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 22 (39)
Lymphopenia (Blood and lymphatic system disorders) | 2 (5)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (1)
Middle ear/hearing (Ear and labyrinth disorders) | 1 (1)
Mood alteration-anxiety, agitation (Psychiatric disorders) | 9 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Nausea (General disorders) | 31 (70)
Neuropathy-sensory (Nervous system disorders) | 10 (11)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 23 (38)
Pain (General disorders) | 10 (12)
Pain-Other (specify, pelvic) (General disorders) | 9 (11)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 3 (3)
Platelets (Blood and lymphatic system disorders) | 11 (13)
Proctitis (Gastrointestinal disorders) | 11 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Radiation Dermatitis (Injury, poisoning and procedural complications) | 6 (8)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10 (15)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 11 (12)
Rectal or perirectal pain (proctalgia) (General disorders) | 6 (9)
Rigors, chills (General disorders) | 27 (46)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 17 (25)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 21 (34)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Stomatitis/pharyngitis (ora/pharyngeal mucositis) (Gastrointestinal disorders) | 5 (6)
Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Vaginal bleeding (Reproductive system and breast disorders) | 20 (34)
Vomiting (Gastrointestinal disorders) | 21 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes